CLINICAL TRIAL: NCT06274437
Title: A Phase 1, Dose Escalation and Dose Optimization Study of the Safety, Tolerability, and Anti-tumor Activity of BND-35 Administered Alone and in Combination With Nivolumab or With Cetuximab in Patients With Advanced Solid Tumors
Brief Title: A Study of BND-35 in Participants With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Biond Biologics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BND-35-001
Record Dates: First submitted 2024-02-14; First posted 2024-02-23 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Antibodies, Monoclonal; Nivolumab; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- BND-35 Dose Escalation (Sub-Part 1A) (Experimental): Accelerated titration followed by standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. BND-35 will be administered at escalating doses of 0.3 mg/kg to 20 mg/kg intravenously (IV), every 2 weeks (Q2W)
  Interventions: Drug: BND-35
- BND-35 in Combination with Nivolumab Dose Escalation (Sub-Part 1B) (Experimental): Standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. BND-35 will be administered at escalating doses of 3 mg/kg to 20 mg/kg intravenously (IV) every 2 weeks (Q2W). Nivolumab will be administered at a dose of 240 mg IV, every 2 weeks (Q2W).
  Interventions: Drug: BND-35; Drug: Nivolumab
- BND-35 in Combination with Cetuximab Dose Escalation (Sub-Part 1C) (Experimental): Standard "3 + 3" dose escalation design with enrollment of at least 3 participants per dose level cohort. BND-35 will be administered at escalating doses of 3 mg/kg to 20 mg/kg intravenously (IV) every 2 weeks (Q2W). Cetuximab will be administered intravenously (IV) at a dose of 500 mg/m2, every 2 weeks (Q2W)
  Interventions: Drug: BND-35; Drug: Cetuximab
- BND-35 in Combination with Nivolumab Dose Optimization (Sub-Part 2A) (Experimental): BND-35 dose optimization in combination with nivolumab. The indications for the combination cohorts will be selected following completion of Part 1. Enrollment will start after the recommended dose(s) of BND-35 have been determined based on data from Sub-Parts 1A, 1B, and 1C. Nivolumab will be administered at a dose of 240 mg IV, every 2 weeks (Q2W).
  Interventions: Drug: BND-35; Drug: Nivolumab
- BND-35 in Combination with Cetuximab Dose Optimization (Sub-Part 2B) (Experimental): BND-35 dose optimization in combination with cetuximab. The indications for the combination cohorts will be selected following completion of Part 1. Enrollment will start after the recommended dose(s) of BND-35 have been determined based on data from Sub-Parts 1A, 1B, and 1C. Cetuximab will be administered intravenously (IV) at a dose of 500 mg/m2, every 2 weeks (Q2W)
  Interventions: Drug: BND-35; Drug: Cetuximab

INTERVENTIONS:
Drug: BND-35 — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: Monoclonal antibody
Drug: Nivolumab — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: Opdivo
  Arms: BND-35 in Combination with Nivolumab Dose Escalation (Sub-Part 1B); BND-35 in Combination with Nivolumab Dose Optimization (Sub-Part 2A)
Drug: Cetuximab — Pharmaceutical form: Solution for infusion; Route of administration: Intravenous
  Other Names: Erbitux
  Arms: BND-35 in Combination with Cetuximab Dose Escalation (Sub-Part 1C); BND-35 in Combination with Cetuximab Dose Optimization (Sub-Part 2B)

SUMMARY:
This is an open-label, multicenter, dose escalation and dose optimization study designed to evaluate safety, tolerability and preliminary anti-tumor activity of BND-35 administered alone and in combination with nivolumab or with cetuximab. The study will enroll advanced cancer patients with unresectable or metastatic disease who are refractory to or are not candidates for standard approved therapy. The study will be comprised of two parts - a dose escalation phase (Part 1) and a dose optimization (Part 2). Part 1 is comprised of three sub-parts: BND-35 administered alone (Sub-Part 1A), BND-35 administered in combination with nivolumab (Sub-Part 1B), and BND-35 administered in combination with cetuximab (Sub-Part 1C). Part 2 is composed of two sub-parts: a dose optimization part where up to two doses of BND-35 per indication are administered in combination with nivolumab or with cetuximab.

DETAILED DESCRIPTION:
Estimated Study Duration:

Dose Escalation (Part 1): Approximately 34 months. Dose Optimization/Expansion (Part 2): Approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unresectable or metastatic disease who are refractory to or are not candidates for standard approved therapy
* Histologic confirmation of malignancy
* Measurable disease per RECIST v1.1
* Eastern Cooperative Oncology Group Performance Status (ECOG) of 0 or 1
* Participants must have adequate organ function as defined by laboratory tests
* Part 1: Following tumor types: Breast cancer, cholangiocarcinoma, colorectal cancer, adenocarcinoma or squamous cell carcinoma of the esophagus, gastric or gastroesophageal junction adenocarcinoma, squamous cell carcinoma of the head and neck, non-small cell lung cancer, melanoma, ovarian cancer, renal cell carcinoma, pancreatic adenocarcinoma, soft tissue sarcomas

Exclusion Criteria:

* Active, known or suspected autoimmune disease
* Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications
* Brain or leptomeningeal metastases
* Known history of positive test for HIV or known AIDS
* Acute or chronic hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Participants after solid organ or allogeneic hematopoietic stem cell transplant
* History of life-threatening toxicity related to prior immune therapy
* History of life-threatening toxicity related to prior cetuximab or other anti-epidermal growth factor receptor antibodies (for Sub-Part 1C)
* Unstable or deteriorating cardiovascular disease within the previous 6 months
* Any major surgery within 4 weeks of study drug administration
* Prior immune therapy treatments, unless at least 4 weeks have elapsed from last dose
* Cytotoxic/Non-cytotoxic anti-cancer agents, unless at least 4 weeks have elapsed from last dose
* Use of other investigational drugs within 28 days
* Prior treatment with immunoglobulin-like transcripts (ILT3)-targeting agents
* Administration of a live attenuated vaccine within 28 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2024-06-02 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Part 1: Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | Through study completion, up to approximately 34 months
  Adverse event (AE): any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of study drug, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent events were events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state up to 30 days after last administration. TEAEs included both Serious TEAEs and non-serious TEAEs.
Part 1: Proportion of patients who discontinued study treatment due to TEAEs | Through study completion, up to approximately 34 months
  Number of patients who discontinued study treatment due to TEAEs
Part 1: Incidence of TEAEs dose limiting toxicities (DLT) | Up to 21 days in Cycle 1
  Incidence of TEAEs meeting protocol defined DLT criteria
Part 2: Objective Response Rate (ORR) per RECIST v1.1 | Through study completion, up to approximately 24 months
  Proportion of participants with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1
Part 2: Incidence of TEAEs and SAEs | Through study completion, an average of 24 months
  Adverse event (AE): any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of study drug, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent events were events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state up to 30 days after last administration. TEAEs included both Serious TEAEs and non-serious TEAEs.

SECONDARY OUTCOMES:
Part 1: Objective Response Rate (ORR) per RECIST v1.1 | Through study completion, up to approximately 34 months
  Proportion of participants with a best overall response of complete response (CR) or partial response (PR) per RECIST v1.1
Part 1: Maximum observed plasma concentration (Cmax) | Through study completion, up to approximately 34 months
  Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Part 1: Serum concentration at the end of the dosing interval (Ctrough) | Through study completion, up to approximately 34 months
  Ctrough is the lowest concentration of drug reached before the next dose was administered.
Part 1: Time of maximum observed serum concentration (Tmax) | Through study completion, up to approximately 34 months
  Tmax is time to reach maximum observed serum concentration obtained directly from the concentration versus time curve.
Part 1: Terminal elimination half-life (T1/2) | Through study completion, up to approximately 34 months
  Terminal half-life is the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination.
Part 1: Area under the plasma concentration-time curve (AUC) | Through study completion, up to approximately 34 months
  AUC is the area under the concentration-time curve of drug
Part 1: Incidence of anti-drug antibodies (ADA) | Through study completion, up to approximately 34 months
  Number of participants with ADA positive results for BND-35
Part 2: Progression Free Survival (PFS) | Through study completion, up to approximately 24 months
  PFS is the time from the date of first dose of study drug to the date of first documented disease progression or death due to any cause, whichever occurs first.
Part 2: PFS rate | At 3, 6, 9, and 12 months, and up to 24 months
  Percentage of participants with PFS, per RECIST v1.1
Part 2: Duration of Response | Through study completion, up to approximately 24 months
  Duration between first documentation of CR or PR to first documentation of disease progression or death due to any cause, whichever occurs first
Part 2: Maximum observed plasma concentration (Cmax) | Through study completion, up to approximately 24 months
  Cmax is the maximum observed serum concentration obtained directly from the concentration versus time curve.
Part 2: Serum concentration at the end of the dosing interval (Ctrough) | Through study completion, up to approximately 24 months
  Ctrough is the lowest concentration of drug reached before the next dose was administered.
Part 2: Time of maximum observed serum concentration (Tmax) | Through study completion, up to approximately 24 months
  Tmax is time to reach maximum observed serum concentration obtained directly from the concentration versus time curve.
Part 2: Terminal elimination half-life (T1/2) | Through study completion, up to approximately 24 months
  Terminal half-life is the time required for the serum concentration of drug to decrease 50 percent in the final stage of its elimination.
Part 2: Area under the plasma concentration-time curve (AUC) | Through study completion, up to approximately 24 months
  AUC is the area under the concentration-time curve of drug
Part 2: Incidence of anti-drug antibodies (ADA) | Through study completion, up to approximately 24 months
  Number of participants with ADA positive results for BND-35

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Ashtamker, Study Director — Biond Bio
Locations (5):
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah University Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv

IPD SHARING:
Plan to Share IPD: No